CLINICAL TRIAL: NCT07136675
Title: Healthy Adult Reference Biobank for Cardiovascular Biomarkers in China
Acronym: HARBOR
Status: Enrolling by invitation | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: HARBOR Study
Record Dates: First submitted 2025-08-13; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy Individuals (Controls)
Keywords: Healthy population, high-sensitivity troponin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Establishing reference intervals for high-sensitivity cardiac troponin in the apparently healthy population in China.

DETAILED DESCRIPTION:
This study was led by Fuwai Hospital, Chinese Academy of Medical Sciences, and implemented as an observational clinical study in collaboration with multiple centers. It selected residual blood samples from individuals who had undergone physical examinations, had signed informed consent, and had no significant abnormalities in routine laboratory tests. High-sensitivity cardiac troponin was measured to establish reference intervals for cardiovascular biomarkers in the apparently healthy population in China.

ELIGIBILITY:
Inclusion criteria:

Apparent healthy Chinese individuals, aged between 20 and 80 years; Normal electrocardiogram (ECG) during physical examination; Signed informed consent form.

Exclusion criteria:

Musculoskeletal disease or a history of rheumatoid arthritis, or high-intensity exercise (e.g., marathon) within the past week; Biotin treatment within the past week; Hospitalization for an emergency within the past three months; Pregnancy or lactation within the past year; Diabetes: fasting blood glucose ≥ 7.0 mmol/L; glycated hemoglobin (HbA1c) ≥ 6.5%; Chronic kidney disease: estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m²; Latent heart disease: NT-proBNP > 125 ng/L or BNP > 35 ng/L; Known cardiovascular or heart disease in the past: treated with medication or other interventions; Chronic diseases that may affect the heart (cancer/tumor, autoimmune diseases); Hemolysis, lipemia, or insufficient residual sample volume for testing.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy population
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Detection of high-sensitivity troponin | On the day of the physical examination
  High-sensitivity troponin, establishment of reference intervals

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No